CLINICAL TRIAL: NCT06696105
Title: Clinical and Laboratory Evaluation of Icon® Resin Infiltration and Vanish™ XT Varnish, on Color Changes of White Spot Lesions
Brief Title: Assessing the Effects of Resin Infiltration and Resin Modified Glass Ionomer on the Color Changes of White Spot Lesions in a Clinical and Laboratory Setting
Acronym: RI
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Deem Abdullah Al-Blaihed, Principal Investigator, King Abdulaziz University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 140-07-23
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: White Spot Lesions; White Spot Lesions [Initial Caries] on Smooth Surface of Tooth; Enamel Hypomineralization
Keywords: "camouflage", "prevention", white spot lesion", "remineralization"
MeSH Terms: conditions — Dental Enamel Hypomineralization

STUDY DESIGN:
Intervention Model Description: the lesions will receive restorative minimally invasive treatment
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Resin infiltration arm (Experimental): resin infiltration will be applied on white spot lesion of anterior teeth
  Interventions: Drug: Resin infiltration
- vanish xt varnish arm (Experimental): vanish xt will be applied on white spot lesion of anterior teeth
  Interventions: Drug: Vanish XT varnish (resin modified glass ionomer restoration)

INTERVENTIONS:
Drug: Resin infiltration — "Icon® resin infiltration (DMG America, Englewood, NJ, US)" technique utilizes light-cured hydrophilic and low viscosity resins that can permeate WSL subsurface micropores. Resin modified glass ionomer cement includes Fluoroaluminosilicate glass, which facilitates the interaction of fluoride with the enamel surface resulting in an instant release . Concurrently, the predominant glass matrix serves as source of fluoride for the purpose of continuous release, hypothesized to facilitate remineralization.
  Other Names: RI
  Arms: Resin infiltration arm
Drug: Vanish XT varnish (resin modified glass ionomer restoration) — Resin modified glass ionomer cement includes Fluoroaluminosilicate glass, which facilitates the interaction of fluoride with the enamel surface resulting in an instant release. Concurrently, the predominant glass matrix serves as source of fluoride for the purpose of continuous release, hypothesized to facilitate remineralization.
  Other Names: Vanish XT varnish
  Arms: vanish xt varnish arm

SUMMARY:
The goal of this clinical trial is to assess the efficacy of "Icon® resin infiltration" and "VanishTM XT varnish" in restoring the appearance of white spot lesions WSLs in healthy children affected with anterior white spot lesions. The main questions it aims to answer are:

1- Are Icon resin infiltration (RI) and Vanish™ XT varnish comparable in restoring esthetics of white spot lesions? Researchers will compare Resin infiltration to vanish xt varnish to see if they are effective in masking white spot lesions

Participants will:

* Have their white spot lesions treated in the dental clinic by the intervention methods
* Visit the clinic after 1 month, 3 months and 6 months to assess the restorations objectively and subjectively

DETAILED DESCRIPTION:
Aim

1. Clinically assess the efficacy of "Icon® resin infiltration" and "VanishTM XT varnish" in restoring the appearance of WSLs
2. Assess patients/parents' satisfaction after "Icon® resin infiltration" and VanishTM XT varnish" application.
3. Evaluate the changes in lesion size by using cross-polarization photography. Materials and Methods The study will be carried out in the "Department of Pediatric Dentistry, Faculty of Dentistry, King Abdulaziz University (KAU)", after approval from the Research Ethics Committee.

Study design A randomized, controlled trial comparing the application of "Icon® resin infiltration" and "VanishTM XT varnish" in parallel groups with a 1:1 allocation ratio. Also, an experimental in vitro study will be conducted.

Clinical trial (Color measurement) Participants, eligibility criteria, and settings A convenient sample of participants attending "King Abdulaziz University Dental Hospital" "KAUDH" will be recruited with WSLs affecting at least one of the labial surfaces of their permanent anterior teeth.

WSLs will be objectively screened Using "DIAGNOdent®" which will quantitively evaluate the loss of the associated fluorescence of WSLs (Q) as well as sound enamel surrounding lesion. The "DIAGNOdent®" device employs blue laser light to illuminate the teeth. The dentin of a tooth comprises fluorophores, which exhibit green fluorescence upon exposure to blue laser light. The presence of a WSL will appear as a dark region surrounded by a green reflective hue, which is observed as a reduction in fluorescence. WSL could easily be overlooked with the absence of "DIAGNOdent®". Only WSLs (Q) scores of 2-9 will be included.

Additionally, WSLs will be subjectively be screened for WSLs using "Enamel Decalcification Index (EDI) by Banks and Richmond" ; only mild and moderate lesions will be considered (level 1 and level 2).

Description of the "EDI by Banks and Richmond" to measure the intensity of White Spot Lesions:

Level 0 = tooth surface without decalcification. Level 1 = clinically visible decalcification of <50% of the examined surface.

Level 2 = moderate to grave decalcification of > 50% of the examined surface.

Level 3 = decalcification on the entire examined surface or cavity, cracking the surface.

As for MIH lesions, criteria of selection will be established according to the European Academy of Pediatric Dentistry (EAPD) policy document. Any lesion with demarcated enamel opacities without a breakdown of the enamel, and induced sensitivity to external stimuli e.g. air/water but not brushing and mild aesthetic concerns on discoloration will be included in the study.

Oral hygiene status The patient's oral hygiene status will be carefully assessed via "Oral Hygiene Index scores by Green and Vermilion" before and during the study period.

Inclusion criteria Exclusion criteria Healthy children aged 6-18 years Any systemic or local conditions not permitting intervention The presence of maxillary permanent anterior teeth. Unwillingness to participate in the study

The finding of a minimum of two white spot lesions (WSLs) on the labial surfaces of maxillary anterior teeth Teeth with periodontal diseases, dental caries, direct or indirect restorations Vital pulp in the anterior teeth. Yellow-brownish opacities with post eruptive enamel breakdown

Patients' enrollment Informed consent forms will be obtained from the parents/guardians for the child's participation in the research.

Sample size calculation The sample size for the clinical trial was determined using "G power software". A significance level of 0.05 and a power of 85% was used as a base for calculations. The outcome will be the variance in color as well as the fluorescence values between treatment groups over a period of three to six months. It is estimated that 88 WSL (44 WSL in each arm), would be adequate.

Randomization In order to achieve even allocation of intervention modalities, computer-generated software available at www.randomization.com will be utilized. The program will employ a block allocation sequence consisting of the following patterns: "AABB, ABBA, BBAA, and BAAB." Group A- will include "icon® resin infiltration", Group B will include "Vanish™ XT varnish".

Allocation concealment and blinding of participants The patients will be blinded to the intervention procedures. The implementation of additional blinding measures will not be feasible due to the variations in material application procedures employed by the intervention approaches. Concealment of the boxes of the material will be done to ensure patients blinding. The same clinician will perform all the procedures.

Intervention methods

Group A: "Icon® resin infiltration" (n=44 teeth):

First, "Icon® Etch, DMG" will be spread for 2 minutes on the tooth affected with WSLs. Following this, water will be used to rinse, then air blowing. Afterwards, the application of "Icon® Dry, DMG" will be done for 30 seconds, followed by air blowing. The "Icon® Infiltrant, DMG" will be spread with the provided sponge applicator and left for three minutes to allow infiltration, then it will be followed by light curing for about sixty seconds.

Group B: "Vanish™ XT varnish" (n=44 teeth):

First, "37% orthophosphoric acid gel" will be applied on the WSL for 15 seconds. Then the paste and liquid components will be mixed on a paper pad for fifteen seconds via an agate spatula, then it will be spread on the WSLs. The material will then be lighted cured for twenty seconds.

Color measurement Both the treatment techniques will be evaluated using the "VITA Easyshade® advance spectrophotometer" before intervention as a baseline reading (T0), then right after intervention (T1), then three months later (T2), then six months later (T3). Photographs will be recorded at every interval. At (T0), the mapping of the dimensions and location of WSL will be done to assess the size and location of the WSLs to ensure an accurate reading.

Size determination using cross-polarisation photography A cross-polarisation filter suitable for our camera (Marumi, Japan) will be used before obtaining the intraoral photographs to minimize light reflection and glare and to be able to observe the lesion borders more clearly. Using photo retractors, intraoral photographs of the treatment and control groups will be obtained before; immediately after; and 1, 3 months after the application of the intervention methods. Next, these images will be analyzed using Image J (1.31o, National Institutes of Health, Bethesda, MD, USA) software, and the lesion areas of the teeth in the treatment group will be measured in mm. The differences in the measurements will be compared with each other at every interval to assess the size of the lesion.

Questionnaire of patients/parents' satisfaction after "Icon resin infiltration" and "Vanish™ XT varnish" application Questionnaires filled out by patients/parents assessing the comfort, complexity, time, and difficulties during the implementation of the intervention strategies. The first section of the questionnaire pertains to the child's demographic information, specifically their name, age and gender. The second section of the questionnaire includes 12 multiple choice questions about the dental restoration's over-all satisfaction, longevity, sensitivity, color, texture and associated defects.

ELIGIBILITY:
Inclusion criteria

* Healthy children
* Presence of maxillary permanent anterior teeth with white spot lesions
* Vital pulp in the anterior teeth.

Exclusion Criteria:

* Any systemic or local conditions not permitting intervention
* Unwillingness to participate in the study
* Teeth with periodontal diseases, dental caries, direct or indirect restorations, yellow-brownish opacities with post eruptive enamel breakdown.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
color measurement | 6 months
  The variance in the value of colors that are observed between two cohorts undergoing therapy, using vita shade spectrophotometer over a six-month period.

SECONDARY OUTCOMES:
color stability | 6 months
  The stability of the colors of the two intervention techniques using vita shade spectrophotometer.

CONTACTS AND LOCATIONS:
Overall Officials: Omar El-Meligy, MSc,Ph.D., Study Director — King Abdulaziz University
Locations (2):
- Saudi Arabia (2):
  - King Abdulaziz University, Jeddah, Saudi Arabia
  - King Abdulaziz University, Jeddah

IPD SHARING:
Plan to Share IPD: No
Data is a part of a thesis and will be published through the research team only

REFERENCES:
- [Background] Al-Haj Ali SN, Alsulaim HN, Albarrak MI, Farah RI. Spectrophotometric comparison of color stability of microhybrid and nanocomposites following exposure to common soft drinks among adolescents: an in vitro study. Eur Arch Paediatr Dent. 2021 Aug;22(4):675-683. doi: 10.1007/s40368-021-00605-6. Epub 2021 Feb 10. PMID 33566286
- [Background] Wiewiora C, Armbruster P, Lallier T, Ballard R. Effectiveness of Vanish XT in Reducing the Development of White Spot Lesions: An In Vitro Study. Oral Health Prev Dent. 2018;16(4):345-350. doi: 10.3290/j.ohpd.a40938. PMID 30175332
- [Background] Kannan A, Padmanabhan S. Comparative evaluation of Icon(R) resin infiltration and Clinpro XT varnish on colour and fluorescence changes of white spot lesions: a randomized controlled trial. Prog Orthod. 2019 Jun 17;20(1):23. doi: 10.1186/s40510-019-0276-y. PMID 31204437
- [Background] Giray FE, Durhan MA, Haznedaroglu E, Durmus B, Kalyoncu IO, Tanboga I. Resin infiltration technique and fluoride varnish on white spot lesions in children: Preliminary findings of a randomized clinical trial. Niger J Clin Pract. 2018 Dec;21(12):1564-1569. doi: 10.4103/njcp.njcp_209_18. PMID 30560818
- [Background] Mehta A, Paramshivam G, Chugh VK, Singh S, Halkai S, Kumar S. Effect of light-curable fluoride varnish on enamel demineralization adjacent to orthodontic brackets: an in-vivo study. Am J Orthod Dentofacial Orthop. 2015 Nov;148(5):814-20. doi: 10.1016/j.ajodo.2015.05.022. PMID 26522042